CLINICAL TRIAL: NCT01015118
Title: Multicenter, Randomised, Double-blind Phase III Trial to Investigate the Efficacy and Safety of BIBF 1120 in Combination With Carboplatin and Paclitaxel Compared to Placebo Plus Carboplatin and Paclitaxel in Patients With Advanced Ovarian Cancer
Brief Title: LUME-Ovar 1: Nintedanib (BIBF 1120) or Placebo in Combination With Paclitaxel and Carboplatin in First Line Treatment of Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.15; AGO-OVAR12 (Other: OTHER); 2008-006831-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-11-09; First posted 2009-11-18 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Ovarian Neoplasms; Peritoneal Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms | interventions — Paclitaxel; nintedanib; Carboplatin

ARMS (2):
- BIBF 1120 (Experimental): patients to receive BIBF 1120 standard dose twice daily PO in combination with combination with carboplatin and paclitaxel
  Interventions: Drug: BIBF 1120; Drug: Paclitaxel; Drug: Carboplatin
- Placebo (Placebo Comparator): patients to receive capsules identical to those containing BIBF 1120 in combination with combination with carboplatin and paclitaxel
  Interventions: Drug: Placebo; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Placebo — comparator to BIBF 1120
  Arms: Placebo
Drug: Paclitaxel — Paclitaxel (standard chemo-therapy)
  Arms: Placebo
Drug: BIBF 1120 — comparison of BIBF 1120 in combination with chemotherapy and placebo in combination with chemotherapy (paclitaxel/carboplatin)
  Arms: BIBF 1120
Drug: Carboplatin — Carboplatin (standard chemo-therapy)
  Arms: Placebo
Drug: Paclitaxel — Paclitaxel (standard chemo-therapy)
  Arms: BIBF 1120
Drug: Carboplatin — Carboplatin (standard chemo-therapy)
  Arms: BIBF 1120

SUMMARY:
The trial will be performed to evaluate if BIBF 1120 in combination with paclitaxel and carboplatin is more effective than placebo in combination with paclitaxel and carboplatin in first-line treatment of patients with advanced ovarian cancer. Safety information about BIBF1120/paclitaxel/carboplatin will be obtained.

ELIGIBILITY:
Inclusion criteria:

* first diagnosis of histologically confirmed epithelial ovarian cancer, fallopian tube or primary peritoneal cancer
* International Federation of Gynecology and Obstetrics (FIGO) Stages IIB - IV
* females, age 18 years or older
* life expectancy of at least 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* prior surgery, defined as either (a) debulking surgery with maximum surgical effort at cytoreduction with the goal of no residual disease or (b) biopsy or limited surgery in patients with stage IV disease for whom surgical debulking was not considered appropriate, if diagnosis is confirmed by histology and no surgery is planned prior to disease progression (including interval debulking surgery)
* patient has given written informed consent which must be consistent with the International Conference on Harmonization - Good Clinical Practice (ICH-GCP) and local legislation
* planned application of first dose of chemotherapy after wound healing, but no later than 10 weeks after surgery

Exclusion criteria:

* histologic diagnosis of a benign or borderline tumour or of a malignant tumour of non-epithelial origin of the ovary, the fallopian tube or the peritoneum
* planned surgery within 124 weeks after randomisation in this trial, including interval debulking surgery
* clinically relevant non-healing wound, ulcer or bone fracture
* clinical symptoms or signs of gastrointestinal obstruction that require parenteral nutrition or hydration
* brain metastases
* pre-existing sensory or motor neuropathy Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher, except due to trauma
* history of major thromboembolic event
* known inherited or acquired bleeding disorder
* significant cardiovascular diseases
* clinically relevant pericardial effusion
* history of a cerebral vascular accident, transient ischemic attack or subarachnoid haemorrhage within the past 6 months
* inadequate safety laboratory values
* serious infections in particular if requiring systemic antibiotic (antimicrobial, antifungal) or antiviral therapy, including Hepatitis B, Hepatitis C, Human Immunodeficiency Virus (HIV)
* poorly controlled diabetes mellitus or other contraindication to high dose corticosteroid therapy
* gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
* other malignancy diagnosed within the past 5 years. In exception to this rule, the following malignancies may be included if adequately treated: non-melanomatous skin cancer, cervical carcinoma in situ, carcinoma in situ of the breast, low risk endometrial cancer
* prior systemic therapy for ovarian cancer (e.g. chemotherapy, monoclonal antibody therapy, oral targeted therapy, hormonal therapy)
* prior systemic cytotoxic chemotherapy
* prior treatment with BIBF 1120 or any other angiogenesis inhibitor
* prior radiotherapy
* serious illness or concomitant non-oncological disease such as neurologic, psychiatric or infectious disease or a laboratory abnormality that may increase the risk associated with study participation or study drug administration
* Women of childbearing potential who are sexually active and not using a highly effective method of birth control during the trial and for at least twelve months after the end of active therapy.
* pregnancy or breast feeding
* psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
* active alcohol or drug abuse
* patients unable to comply with the protocol
* any contraindications for therapy with paclitaxel or carboplatin
* treatment with other investigational drugs or participation in another clinical trial testing a drug within the past four weeks before start of therapy or concomitantly with this trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1366 (Actual)
Dates: Start 2009-11-17 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (281):
- United States (33):
  - 1199.15.10113 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 1199.15.10030 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1199.15.10001 Boehringer Ingelheim Investigational Site, Santa Rosa, California
  - 1199.15.10005 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 1199.15.10028 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 1199.15.10014 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1199.15.10010 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 1199.15.10004 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 1199.15.10011 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1199.15.10003 Boehringer Ingelheim Investigational Site, Marrero, Louisiana
  - 1199.15.10017 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1199.15.10103 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1199.15.10002 Boehringer Ingelheim Investigational Site, New York, New York
  - 1199.15.10012 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1199.15.10020 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1199.15.10019 Boehringer Ingelheim Investigational Site, Bismarck, North Dakota
  - 1199.15.10024 Boehringer Ingelheim Investigational Site, Canton, Ohio
  - 1199.15.10025 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 1199.15.10029 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 1199.15.10021 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1199.15.10013 Boehringer Ingelheim Investigational Site, Abington, Pennsylvania
  - 1199.15.10016 Boehringer Ingelheim Investigational Site, Allentown, Pennsylvania
  - 1199.15.10008 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 1199.15.10102 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1199.15.10006 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1199.15.10104 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1199.15.10100 Boehringer Ingelheim Investigational Site, Bedford, Texas
  - 1199.15.10107 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1199.15.10108 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1199.15.10110 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1199.15.10007 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1199.15.10105 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1199.15.10112 Boehringer Ingelheim Investigational Site, Vancouver, Washington
- Australia (7):
  - 1199.15.61006 Boehringer Ingelheim Investigational Site, Camperdown, New South Wales
  - 1199.15.61001 Boehringer Ingelheim Investigational Site, Waratah, New South Wales
  - 1199.15.61004 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 1199.15.61003 Boehringer Ingelheim Investigational Site, Southe Brisbane, Queensland
  - 1199.15.61005 Boehringer Ingelheim Investigational Site, North Terrace, South Australia
  - 1199.15.61007 Boehringer Ingelheim Investigational Site, Parkville, Victoria
  - 1199.15.61002 Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
- Austria (9):
  - 1199.15.43003 Boehringer Ingelheim Investigational Site, Graz
  - 1199.15.43001 Boehringer Ingelheim Investigational Site, Innsbruck
  - 1199.15.43011 Boehringer Ingelheim Investigational Site, Krems
  - 1199.15.43007 Boehringer Ingelheim Investigational Site, Kufstein
  - 1199.15.43005 Boehringer Ingelheim Investigational Site, Linz
  - 1199.15.43010 Boehringer Ingelheim Investigational Site, Salzburg
  - 1199.15.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 1199.15.43012 Boehringer Ingelheim Investigational Site, Vienna
  - 1199.15.43013 Boehringer Ingelheim Investigational Site, Wels
- Belgium (6):
  - 1199.15.32010 Boehringer Ingelheim Investigational Site, Edegem
  - 1199.15.32012 Boehringer Ingelheim Investigational Site, Hasselt
  - 1199.15.32003 Boehringer Ingelheim Investigational Site, La Louvière
  - 1199.15.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 1199.15.32007 Boehringer Ingelheim Investigational Site, Liège
  - 1199.15.32008 Boehringer Ingelheim Investigational Site, Sint-Niklaas
- Canada (7):
  - 1199.15.11005 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1199.15.11004 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1199.15.11008 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1199.15.11009 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1199.15.11003 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1199.15.11006 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1199.15.11001 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- Czechia (3):
  - 1199.15.42002 Boehringer Ingelheim Investigational Site, Brno
  - 1199.15.42003 Boehringer Ingelheim Investigational Site, Olomouc
  - 1199.15.42001 Boehringer Ingelheim Investigational Site, Prague
- Denmark (5):
  - 1199.15.45004 Boehringer Ingelheim Investigational Site, Aalborg
  - 1199.15.45002 Boehringer Ingelheim Investigational Site, Herlev
  - 1199.15.45005 Boehringer Ingelheim Investigational Site, Herning
  - 1199.15.45001 Boehringer Ingelheim Investigational Site, Købenahvn Ø
  - 1199.15.45003 Boehringer Ingelheim Investigational Site, Odense C
- Finland (5):
  - 1199.15.35801 Boehringer Ingelheim Investigational Site, Helsinki
  - 1199.15.35804 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1199.15.35805 Boehringer Ingelheim Investigational Site, Kuopio
  - 1199.15.35803 Boehringer Ingelheim Investigational Site, Oulu
  - 1199.15.35802 Boehringer Ingelheim Investigational Site, Tampere
- France (31):
  - 1199.15.33047 Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - 1199.15.33035 Boehringer Ingelheim Investigational Site, Avignon
  - 1199.15.33055 Boehringer Ingelheim Investigational Site, Besançon
  - 1199.15.33003 Boehringer Ingelheim Investigational Site, Bordeaux
  - 1199.15.33004 Boehringer Ingelheim Investigational Site, Bordeaux
  - 1199.15.33006 Boehringer Ingelheim Investigational Site, Caen
  - 1199.15.33025 Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1199.15.33048 Boehringer Ingelheim Investigational Site, Dechy
  - 1199.15.33042 Boehringer Ingelheim Investigational Site, Fréjus
  - 1199.15.33037 Boehringer Ingelheim Investigational Site, La Roche-sur-Yon
  - 1199.15.33008 Boehringer Ingelheim Investigational Site, Le Mans
  - 1199.15.33009 Boehringer Ingelheim Investigational Site, Lille
  - 1199.15.33020 Boehringer Ingelheim Investigational Site, Lyon
  - 1199.15.33011 Boehringer Ingelheim Investigational Site, Marseille
  - 1199.15.33021 Boehringer Ingelheim Investigational Site, Monaco Cedex
  - 1199.15.33012 Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 1199.15.33052 Boehringer Ingelheim Investigational Site, Montpellier
  - 1199.15.33053 Boehringer Ingelheim Investigational Site, Mougins
  - 1199.15.33038 Boehringer Ingelheim Investigational Site, Nancy
  - 1199.15.33013 Boehringer Ingelheim Investigational Site, Nantes
  - 1199.15.33015 Boehringer Ingelheim Investigational Site, Orléans
  - 1199.15.33001 Boehringer Ingelheim Investigational Site, Paris
  - 1199.15.33027 Boehringer Ingelheim Investigational Site, Paris
  - 1199.15.33051 Boehringer Ingelheim Investigational Site, Périgueux
  - 1199.15.33030 Boehringer Ingelheim Investigational Site, Plerin SUR MER
  - 1199.15.33045 Boehringer Ingelheim Investigational Site, Saint-Cloud
  - 1199.15.33033 Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1199.15.33018 Boehringer Ingelheim Investigational Site, Strasbourg
  - 1199.15.33039 Boehringer Ingelheim Investigational Site, Thonon-les-Bains
  - 1199.15.33031 Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
  - 1199.15.33050 Boehringer Ingelheim Investigational Site, Villejuif
- Germany (78):
  - 1199.15.49040 Boehringer Ingelheim Investigational Site, Aachen
  - 1199.15.49070 Boehringer Ingelheim Investigational Site, Aalen
  - 1199.15.49086 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1199.15.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1199.15.49039 Boehringer Ingelheim Investigational Site, Berlin
  - 1199.15.49041 Boehringer Ingelheim Investigational Site, Berlin
  - 1199.15.49004 Boehringer Ingelheim Investigational Site, Bonn
  - 1199.15.49042 Boehringer Ingelheim Investigational Site, Bonn
  - 1199.15.49071 Boehringer Ingelheim Investigational Site, Bottrop
  - 1199.15.49081 Boehringer Ingelheim Investigational Site, Böblingen
  - 1199.15.49043 Boehringer Ingelheim Investigational Site, Chemnitz
  - 1199.15.49005 Boehringer Ingelheim Investigational Site, Dessau
  - 1199.15.49006 Boehringer Ingelheim Investigational Site, Detmold
  - 1199.15.49007 Boehringer Ingelheim Investigational Site, Dresden
  - 1199.15.49067 Boehringer Ingelheim Investigational Site, Dresden
  - 1199.15.49008 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1199.15.49009 Boehringer Ingelheim Investigational Site, Ebersberg
  - 1199.15.49010 Boehringer Ingelheim Investigational Site, Essen
  - 1199.15.49066 Boehringer Ingelheim Investigational Site, Essen
  - 1199.15.49089 Boehringer Ingelheim Investigational Site, Essen
  - 1199.15.49045 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1199.15.49011 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1199.15.49068 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1199.15.49083 Boehringer Ingelheim Investigational Site, Freudenstadt
  - 1199.15.49046 Boehringer Ingelheim Investigational Site, Fulda
  - 1199.15.49012 Boehringer Ingelheim Investigational Site, Fürstenfeldbruck
  - 1199.15.49064 Boehringer Ingelheim Investigational Site, Greifswald
  - 1199.15.49076 Boehringer Ingelheim Investigational Site, Gütersloh
  - 1199.15.49014 Boehringer Ingelheim Investigational Site, Halle/S.
  - 1199.15.49015 Boehringer Ingelheim Investigational Site, Hamburg
  - 1199.15.49084 Boehringer Ingelheim Investigational Site, Hamburg
  - 1199.15.49073 Boehringer Ingelheim Investigational Site, Hanau
  - 1199.15.49095 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1199.15.49080 Boehringer Ingelheim Investigational Site, Henstedt-Ulzburg
  - 1199.15.49047 Boehringer Ingelheim Investigational Site, Hildesheim
  - 1199.15.49016 Boehringer Ingelheim Investigational Site, Karlsruhe
  - 1199.15.49017 Boehringer Ingelheim Investigational Site, Kiel
  - 1199.15.49062 Boehringer Ingelheim Investigational Site, Krefeld
  - 1199.15.49018 Boehringer Ingelheim Investigational Site, Landshut
  - 1199.15.49087 Boehringer Ingelheim Investigational Site, Ludwigsburg
  - 1199.15.49019 Boehringer Ingelheim Investigational Site, Lübeck
  - 1199.15.49020 Boehringer Ingelheim Investigational Site, Magdeburg
  - 1199.15.49021 Boehringer Ingelheim Investigational Site, Mainz
  - 1199.15.49022 Boehringer Ingelheim Investigational Site, Mainz
  - 1199.15.49023 Boehringer Ingelheim Investigational Site, Mannheim
  - 1199.15.49024 Boehringer Ingelheim Investigational Site, Marburg
  - 1199.15.49025 Boehringer Ingelheim Investigational Site, München
  - 1199.15.49026 Boehringer Ingelheim Investigational Site, München
  - 1199.15.49027 Boehringer Ingelheim Investigational Site, München
  - 1199.15.49048 Boehringer Ingelheim Investigational Site, München
  - 1199.15.49065 Boehringer Ingelheim Investigational Site, Neumarkt in der Oberpfalz
  - 1199.15.49029 Boehringer Ingelheim Investigational Site, Offenbach
  - 1199.15.49082 Boehringer Ingelheim Investigational Site, Paderborn
  - 1199.15.49030 Boehringer Ingelheim Investigational Site, Radebeul
  - 1199.15.49061 Boehringer Ingelheim Investigational Site, Ravensburg
  - 1199.15.49050 Boehringer Ingelheim Investigational Site, Regensburg
  - 1199.15.49051 Boehringer Ingelheim Investigational Site, Rosenheim
  - 1199.15.49052 Boehringer Ingelheim Investigational Site, Rostock
  - 1199.15.49054 Boehringer Ingelheim Investigational Site, Saalfeld
  - 1199.15.49031 Boehringer Ingelheim Investigational Site, Salzgitter
  - 1199.15.49055 Boehringer Ingelheim Investigational Site, Solingen
  - 1199.15.49092 Boehringer Ingelheim Investigational Site, Stadthagen
  - 1199.15.49063 Boehringer Ingelheim Investigational Site, Stendal
  - 1199.15.49093 Boehringer Ingelheim Investigational Site, Stralsund
  - 1199.15.49033 Boehringer Ingelheim Investigational Site, Stuttgart
  - 1199.15.49056 Boehringer Ingelheim Investigational Site, Stuttgart
  - 1199.15.49090 Boehringer Ingelheim Investigational Site, Stuttgart
  - 1199.15.49079 Boehringer Ingelheim Investigational Site, Suhl
  - 1199.15.49034 Boehringer Ingelheim Investigational Site, Traunstein
  - 1199.15.49057 Boehringer Ingelheim Investigational Site, Trier
  - 1199.15.49035 Boehringer Ingelheim Investigational Site, Tübingen
  - 1199.15.49058 Boehringer Ingelheim Investigational Site, Ulm
  - 1199.15.49085 Boehringer Ingelheim Investigational Site, Viersen
  - 1199.15.49001 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 1199.15.49036 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 1199.15.49059 Boehringer Ingelheim Investigational Site, Witten
  - 1199.15.49037 Boehringer Ingelheim Investigational Site, Wolfsburg
  - 1199.15.49060 Boehringer Ingelheim Investigational Site, Worms
- Greece (5):
  - 1199.15.30001 Boehringer Ingelheim Investigational Site, Athens
  - 1199.15.30003 Boehringer Ingelheim Investigational Site, Heraklio
  - 1199.15.30002 Boehringer Ingelheim Investigational Site, Nea Kifissia
  - 1199.15.30005 Boehringer Ingelheim Investigational Site, Pátrai
  - 1199.15.30004 Boehringer Ingelheim Investigational Site, Thessaloniki
- Italy (35):
  - 1199.15.39027 Boehringer Ingelheim Investigational Site, Asti
  - 1199.15.39002 Boehringer Ingelheim Investigational Site, Avellino
  - 1199.15.39003 Boehringer Ingelheim Investigational Site, Aviano (PN)
  - 1199.15.39004 Boehringer Ingelheim Investigational Site, Bari
  - 1199.15.39005 Boehringer Ingelheim Investigational Site, Benevento
  - 1199.15.39029 Boehringer Ingelheim Investigational Site, Brescia
  - 1199.15.39040 Boehringer Ingelheim Investigational Site, Catania
  - 1199.15.39007 Boehringer Ingelheim Investigational Site, Catanzaro
  - 1199.15.39008 Boehringer Ingelheim Investigational Site, Faenza (RA)
  - 1199.15.39039 Boehringer Ingelheim Investigational Site, Ferrara
  - 1199.15.39017 Boehringer Ingelheim Investigational Site, Genova
  - 1199.15.39037 Boehringer Ingelheim Investigational Site, Lecce
  - 1199.15.39009 Boehringer Ingelheim Investigational Site, Mantova
  - 1199.15.39033 Boehringer Ingelheim Investigational Site, Meldola (FC)
  - 1199.15.39021 Boehringer Ingelheim Investigational Site, Milan
  - 1199.15.39028 Boehringer Ingelheim Investigational Site, Milan
  - 1199.15.39036 Boehringer Ingelheim Investigational Site, Milan
  - 1199.15.39010 Boehringer Ingelheim Investigational Site, Modena
  - 1199.15.39026 Boehringer Ingelheim Investigational Site, Monza
  - 1199.15.39001 Boehringer Ingelheim Investigational Site, Napoli
  - 1199.15.39022 Boehringer Ingelheim Investigational Site, Padua
  - 1199.15.39011 Boehringer Ingelheim Investigational Site, Palermo
  - 1199.15.39031 Boehringer Ingelheim Investigational Site, Palermo
  - 1199.15.39023 Boehringer Ingelheim Investigational Site, Pisa
  - 1199.15.39012 Boehringer Ingelheim Investigational Site, Pordenone
  - 1199.15.39024 Boehringer Ingelheim Investigational Site, Reggio Emilia
  - 1199.15.39013 Boehringer Ingelheim Investigational Site, Roma
  - 1199.15.39014 Boehringer Ingelheim Investigational Site, Roma
  - 1199.15.39034 Boehringer Ingelheim Investigational Site, Rozzano (MI)
  - 1199.15.39030 Boehringer Ingelheim Investigational Site, San Fermo della Battaglia
  - 1199.15.39018 Boehringer Ingelheim Investigational Site, Sondrio
  - 1199.15.39006 Boehringer Ingelheim Investigational Site, Tappino (CB)
  - 1199.15.39019 Boehringer Ingelheim Investigational Site, Torino
  - 1199.15.39020 Boehringer Ingelheim Investigational Site, Torino
  - 1199.15.39032 Boehringer Ingelheim Investigational Site, Varese
- Netherlands (6):
  - 1199.15.31009 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1199.15.31005 Boehringer Ingelheim Investigational Site, Amersfoort
  - 1199.15.31004 Boehringer Ingelheim Investigational Site, Niewegein
  - 1199.15.31003 Boehringer Ingelheim Investigational Site, Nijmegen
  - 1199.15.31006 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1199.15.31002 Boehringer Ingelheim Investigational Site, Utrecht
- Norway (4):
  - 1199.15.47003 Boehringer Ingelheim Investigational Site, Bergen
  - 1199.15.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 1199.15.47002 Boehringer Ingelheim Investigational Site, Stavanger
  - 1199.15.47004 Boehringer Ingelheim Investigational Site, Trondheim
- Poland (3):
  - 1199.15.48003 Boehringer Ingelheim Investigational Site, Gdansk
  - 1199.15.48006 Boehringer Ingelheim Investigational Site, Lublin
  - 1199.15.48001 Boehringer Ingelheim Investigational Site, Warsaw
- Portugal (7):
  - 1199.15.35102 Boehringer Ingelheim Investigational Site, Coimbra
  - 1199.15.35104 Boehringer Ingelheim Investigational Site, Coimbra
  - 1199.15.35101 Instituto Portugues de Oncologia Lisboa Francisco Gentil, Lisbon
  - 1199.15.35106 Boehringer Ingelheim Investigational Site, Lisbon
  - 1199.15.35108 Boehringer Ingelheim Investigational Site, Lisbon
  - 1199.15.35105 Boehringer Ingelheim Investigational Site, Porto
  - 1199.15.35109 Boehringer Ingelheim Investigational Site, Vila Real
- Russia (5):
  - 1199.15.70006 Boehringer Ingelheim Investigational Site, Barnaul
  - 1199.15.70007 Boehringer Ingelheim Investigational Site, Kazan'
  - 1199.15.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1199.15.70002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1199.15.70005 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Slovakia (6):
  - 1199.15.42101 Boehringer Ingelheim Investigational Site, Bratislava
  - 1199.15.42105 Boehringer Ingelheim Investigational Site, Bratislava
  - 1199.15.42106 Boehringer Ingelheim Investigational Site, Košice
  - 1199.15.42103 Boehringer Ingelheim Investigational Site, Nitra
  - 1199.15.42104 Boehringer Ingelheim Investigational Site, Poprad
  - 1199.15.42102 Boehringer Ingelheim Investigational Site, Žilina
- Spain (8):
  - 1199.15.34001 Boehringer Ingelheim Investigational Site, Badalona
  - 1199.15.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 1199.15.34006 Boehringer Ingelheim Investigational Site, Girona
  - 1199.15.34004 Boehringer Ingelheim Investigational Site, Lleida
  - 1199.15.34002 Boehringer Ingelheim Investigational Site, Madrid
  - 1199.15.34010 Boehringer Ingelheim Investigational Site, Madrid
  - 1199.15.34005 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1199.15.34009 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (5):
  - 1199.15.46005 Boehringer Ingelheim Investigational Site, Linköping
  - 1199.15.46001 Boehringer Ingelheim Investigational Site, Lund
  - 1199.15.46002 Boehringer Ingelheim Investigational Site, Stockholm
  - 1199.15.46004 Boehringer Ingelheim Investigational Site, Umeå
  - 1199.15.46003 Boehringer Ingelheim Investigational Site, Uppsala
- Ukraine (5):
  - 1199.15.38006 Boehringer Ingelheim Investigational Site, Cherkasy
  - 1199.15.38005 Boehringer Ingelheim Investigational Site, Dnipro
  - 1199.15.38004 Boehringer Ingelheim Investigational Site, Donetsk
  - 1199.15.38002 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1199.15.38003 Boehringer Ingelheim Investigational Site, Lviv
- United Kingdom (8):
  - 1199.15.44006 Boehringer Ingelheim Investigational Site, Derby
  - 1199.15.44007 Boehringer Ingelheim Investigational Site, Dundee
  - 1199.15.44003 Boehringer Ingelheim Investigational Site, Glasgow
  - 1199.15.44001 Boehringer Ingelheim Investigational Site, Guildford
  - 1199.15.44005 Boehringer Ingelheim Investigational Site, London
  - 1199.15.44004 Boehringer Ingelheim Investigational Site, Nottingham
  - 1199.15.44002 Boehringer Ingelheim Investigational Site, Poole
  - 1199.15.44008 Boehringer Ingelheim Investigational Site, Truro

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] du Bois A, Kristensen G, Ray-Coquard I, Reuss A, Pignata S, Colombo N, Denison U, Vergote I, Del Campo JM, Ottevanger P, Heubner M, Minarik T, Sevin E, de Gregorio N, Bidzinski M, Pfisterer J, Malander S, Hilpert F, Mirza MR, Scambia G, Meier W, Nicoletto MO, Bjorge L, Lortholary A, Sailer MO, Merger M, Harter P; AGO Study Group led Gynecologic Cancer Intergroup/European Network of Gynaecologic Oncology Trials Groups Intergroup Consortium. Standard first-line chemotherapy with or without nintedanib for advanced ovarian cancer (AGO-OVAR 12): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet Oncol. 2016 Jan;17(1):78-89. doi: 10.1016/S1470-2045(15)00366-6. Epub 2015 Nov 16. PMID 26590673

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1366 patients were randomised for this study.
Groups:
- Nintedanib: Patients to receive Nintedanib 200 milligram (mg) soft gelatine capsule, taken orally twice daily, except the day of chemotherapy (carboplatin and paclitaxel) infusion, every 21 days for six courses.
- Placebo: Patients to receive matching placebo soft gelatine capsule identical to those containing Nintedanib, taken orally twice daily, except the day of chemotherapy (carboplatin and paclitaxel) infusion, every 21 days for six courses.
Period: Overall Study
Arm/Group | Nintedanib | Placebo
Started | 911 | 455
Completed | 242 (Patients who completed max trial therapy duration.) | 128 (Patients who completed max trial therapy duration.)
Not Completed | 669 | 327
Not completed — Protocol Violation | 5 | 6
Not completed — Withdrawal by Subject | 103 | 27
Not completed — Other Adverse Event (AE) | 141 | 33
Not completed — Worsening or AE of underlying disease | 5 | 4
Not completed — Progressive disease | 364 | 229
Not completed — Not treated | 9 | 5
Not completed — Other than stated above | 42 | 23

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): included all randomised patients, regardless of whether or not they had received treatment. Patients were assigned to nintedanib or placebo as randomised.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib | Placebo | Total
Number analyzed (Participants) | 911 | 455 | 1366
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (11.0) | 56.9 (11.1) | 57.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 911 | 455 | 1366
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PFS Based on Investigator Assessment According to Modified Response Evaluation Criteria in Solid Tumors, Version 1.1 (mRECIST), and Additional Clinical Criteria.
Description: Progression free survival (PFS) is calculated as the time from randomisation to the date of disease progression, or to the date of death, whichever occurs first according to the Investigator assessment.
  The primary PFS analysis of this trial was performed when approximately 753 patients had experienced a PFS event
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve for each treatment arm.
Time Frame: First drug administration to date of disease progression or death whichever occurs first , upto 29 months
Population: Randomised Set (RS)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
Months | 17.2 [11.1 to 32.5] | 16.6 [10.8 to 30.4]
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; Hazard ratio (HR), Confidence Interval (CI) and P-value obtained from a proportional-hazards model stratified by Macroscopic residual postoperative tumour (Yes vs. no), the International Federation of Gynecology and Obstetrics (FIGO) Stage (IIB-III vs. IV) and carboplatin level Area under curve 5 (AUC5) vs. Area under curve 6 (AUC6); Test type: Superiority or Other; p = 0.0239, Log Rank; Breslow method was used for handling ties; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.72 to 0.98] — If hazard ratio is below 1 then favours nintedanib

2. Primary Outcome: PFS Based on Investigator Assessment According to Modified Response Evaluation Criteria in Solid Tumors, Version 1.1 (mRECIST), and Additional Clinical Criteria (Follow up Analysis).
Description: Follow-up analysis was conducted at the time of overall survival analysis. Progression free survival (PFS) is calculated as the time from randomisation to the date of disease progression, or to the date of death, whichever occurs first according to the Investigator assessment.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve for each treatment arm.
Time Frame: First drug administration to date of disease progression or death whichever occurs first until final Data Base Lock (DBL) 26September16, upto 62 months
Population: Randomised Set (RS)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
Months | 17.6 [11.1 to 38.0] | 16.6 [10.8 to 37.3]
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; Hazard ratio (HR), Confidence Interval (CI) and P-value obtained from a proportional-hazards model stratified by Macroscopic residual postoperative tumour (Yes vs. no), the International Federation of Gynecology and Obstetrics (FIGO) Stage (IIB-III vs. IV) and carboplatin level (AUC5 vs. AUC6); Test type: Superiority or Other; p = 0.0286, Log Rank; Breslow method was used for handling ties; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.75 to 0.98] — If hazard ratio is below 1 then favours nintedanib

3. Secondary Outcome: PFS Based on Investigator Assessment According to mRECIST Version 1.1 (Key Secondary Endpoint).
Description: Progression free survival is calculated as the time from randomisation to the date of disease progression, or to the date of death, whichever occurs first based on the Investigator assessment according to Modified Response Evaluation Criteria (mRECIST), version 1.1.
  The primary PFS analysis of this trial was performed when approximately 753 patients had experienced a PFS event.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve for each treatment arm.
Time Frame: First drug administration to date of disease progression or death whichever occurs first , upto 29 months
Population: Randomised Set (RS)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
Months | 18.3 [11.1 to 32.5] | 16.6 [10.8 to 30.4]
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; HR, CI and P-value obtained from a proportional-hazards model stratified by Macroscopic residual postoperative tumour (Yes vs. no), the International Federation of Gynecology and Obstetrics (FIGO) Stage (IIB-III vs. IV) and carboplatin level (AUC5 vs. AUC6); Test type: Superiority or Other; p = 0.0186, Log Rank; Breslow method was used for handling ties; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.72 to 0.97] — If hazard ratio is below 1 then favours nintedanib

4. Secondary Outcome: PFS Based on Investigator Assessment According to mRECIST Version 1.1 (Key Secondary Endpoint - Follow up Analysis).
Description: Follow-up analysis was conducted at the time of overall survival analysis. Progression free survival is calculated as the time from randomisation to the date of disease progression, or to the date of death, whichever occurs first based on the Investigator assessment according to Modified Response Evaluation Criteria (mRECIST), version 1.1. Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve for each treatment arm.
Time Frame: as for outcome 2
Population: Randomised Set (RS)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
Months | 18.4 [11.1 to 38.5] | 16.6 [10.8 to 37.3]
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0256, Log Rank; Breslow method was used for handling ties; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.74 to 0.98] — If hazard ratio is below 1 then favours nintedanib

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from randomization to date of death (irrespective of reason).
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve for each treatment arm.
Time Frame: First drug administration to date of death until final DBL 26September16, upto 62 months
Population: Randomised Set (RS)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
Months | 62.0 [30.0 to NA] — Not calculable because of insufficient number of participants with events | 62.8 [30.6 to NA] — Not calculable because of insufficient number of participants with events
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8653, Log Rank; Breslow method was used for handling ties; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.83 to 1.17] — If hazard ratio is below 1 then favours nintedanib

6. Secondary Outcome: Time to CA-125 Tumour Marker Progression
Description: Time to tumour-marker progression was defined as the time from randomisation until the date when Carbohydrate (cancer) antigen (CA-125) values increased to higher than twice the nadir value. CA-125 >=2 x nadir in case nadir value > Upper limit of normal (ULN) or CA-125 >=2 x ULN in case nadir value <= ULN.
Time Frame: First drug administration until final DBL 26September16, upto 62 months
Population: Randomised set (RS)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
Months | 16.6 [10.6 to 47.0] | 14.1 [8.6 to 42.6]
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0749, Log Rank; Breslow method was used for handling ties; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.77 to 1.01] — If hazard ratio is below 1 then favours nintedanib

7. Secondary Outcome: Objective Response Based on Investigator Assessment
Description: Objective tumour response defined as either complete response [CR] or partial response [PR] in patients with at least 1 target lesion reported at baseline
Time Frame: First drug administration until final DBL 26September16, upto 62 months
Population: Randomised Set (RS) for patients with at least 1 target lesion reported at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
percentage of participants | 74.3 | 70.2
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; Odds ratio and p-value are obtained from logistic regression model adjusting for, macroscopic residual postoperative tumour (yes vs. no), the International Federation of Gynecology and Obstetrics (FIGO) stage (IIB-III vs. IV) and carboplatin level (AUC5 vs. AUC6); Test type: Superiority or Other; p = 0.3490, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.81 to 1.82] — An odds ratio >1 favours nintedanib

8. Secondary Outcome: Change in Abdominal/Gastro-intestinal Symptoms Over Time
Description: Change in abdominal/gastro-intestinal over time was calculated on symptoms (scale composite of items 31 to 37 of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Module for Ovarian Cancer 28 (EORTC QLQ OV-28).
  As specified in the EORTC scoring manual, for each scale or item, a linear transformation was applied to standardize the raw score to a range from 0 to 100 (high scores represent a high/severe level of symptomatology).
  Mean presented is Adjusted mean. Adjusted for the stratification factors macroscopic residual postoperative tumour at baseline (yes vs. no), FIGO stage (IIB-III vs IV), and Carboplatin level (AUC5 vs. AUC6).
Time Frame: First drug administration until final DBL 26September16, upto 62 months
Population: Randomised Set (RS) for patients with abdominal/gastro-intestinal symptoms
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
units on a scale | 24.63 (0.49) | 19.34 (0.64)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; Adjusted for the stratification factors macroscopic residual postoperative tumour at baseline (yes vs. no), the International Federation of Gynecology and Obstetrics (FIGO) stage (IIB-III vs IV), and carboplatin level (AUC5 vs. AUC6); Test type: Superiority or Other; p < 0.0001, Mixed effect growth curve model; Mixed-effects growth curve models (longitudinal models) with the average profile over time for each endpoint described by a piecewise linear model; Mean Difference (Net) = 5.29, 95% CI 2-sided [3.88 to 6.69], Standard Error of Mean 0.72 — Mean difference presented is the Adjusted mean difference. Difference calculated as nintedanib minus placebo. High values represent a worse level of symptoms

9. Secondary Outcome: Change in Global Health Status/ Quality of Life (QoL) Scale Over Time.
Description: Change in Global Health Status/ Quality of life (QoL) over time was calculated on Global Health Status/QoL scale (composite of items 29 and 30 of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-30 (EORTC QLQ-C30) as a general measure.
  As specified in the EORTC scoring manual, for each scale or item, a linear transformation was applied to standardize the raw score to a range from 0 to 100 (high scores represent a high/healthy level of functioning).
  Mean presented is Adjusted mean. Adjusted for the stratification factors macroscopic residual postoperative tumour at baseline (yes vs. no), FIGO stage (IIB-III vs IV), and Carboplatin level (AUC5 vs. AUC6).
Time Frame: First drug administration until final DBL 26September16, upto 62 months
Population: Randomised Set (RS) for patients with global health status/QoL
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 911 | 455
units on a scale | 68.79 (0.48) | 70.67 (0.65)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0124, Mixed effect growth curve model; [statistical method as in outcome 8, analysis 1]; Mean Difference (Net) = -1.88, 95% CI 2-sided [-3.35 to -0.41], Standard Error of Mean 0.75 — Mean difference calculated is the Adjusted mean. High values represent a better level of functioning. Difference calculated as nintedanib minus placebo

ADVERSE EVENTS:
Time Frame: First drug administration until data cut-off 26September16, up to 62 months
Description: Adverse Events were reported for the treated patients.
Arm/Group | Placebo | Nintedanib
Serious Adverse Events (participants affected / at risk) | 157/450 | 379/902
Other Adverse Events (participants affected / at risk) | 442/450 | 891/902
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=450) | Nintedanib (N=902)
Anaemia (Blood and lymphatic system disorders) | 9 | 36
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 20
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 8
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 24
Pancytopenia (Blood and lymphatic system disorders) | 1 | 8
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 21
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Cancer gene carrier (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Goitre (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 30
Abdominal pain upper (Gastrointestinal disorders) | 0 | 8
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 8 | 14
Colitis (Gastrointestinal disorders) | 2 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 10 | 13
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 41
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 2
Faecaloma (Gastrointestinal disorders) | 1 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Fistula of small intestine (Gastrointestinal disorders) | 0 | 2
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 8 | 17
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 7
Intestinal perforation (Gastrointestinal disorders) | 1 | 5
Intussusception (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 10 | 24
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 12
Small intestinal perforation (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 2 | 8
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 12 | 33
Asthenia (General disorders) | 2 | 13
Catheter site haematoma (General disorders) | 1 | 0
Chest pain (General disorders) | 4 | 4
Chills (General disorders) | 0 | 1
Cyst (General disorders) | 1 | 0
Death (General disorders) | 0 | 2
Fatigue (General disorders) | 2 | 10
General physical health deterioration (General disorders) | 5 | 17
Hernia (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Implant site erythema (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 2
Infusion site extravasation (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Nodule (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 2 | 1
Performance status decreased (General disorders) | 1 | 1
Pyrexia (General disorders) | 8 | 23
Sudden death (General disorders) | 2 | 0
Surgical failure (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 4
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 2
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 3 | 9
Hypersensitivity (Immune system disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 2
Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 0 | 6
Device related infection (Infections and infestations) | 3 | 4
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 4
Gastrointestinal infection (Infections and infestations) | 0 | 2
Infected lymphocele (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 3
Infectious pleural effusion (Infections and infestations) | 0 | 1
Joint abscess (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 2
Mesenteric abscess (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 2
Pelvic abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 2
Pharyngeal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 6
Postoperative abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 2
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 4
Septic shock (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 17
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 2
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 2
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 4 | 8
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Biopsy vulva (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 0 | 2
C-reactive protein increased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 3
Electrocardiogram abnormal (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Glomerular filtration rate decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 3
Lipase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 0 | 5
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 3
White blood cell count decreased (Investigations) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 6 | 21
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal wall neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 15
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to reproductive organ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Asterixis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 5
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 5
Hemianopia homonymous (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 6
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Thrombosis in device (Product Issues) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Conversion disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 3
Hallucination (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 4
Bladder tamponade (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 7
Incontinence (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 4
Ureteric obstruction (Renal and urinary disorders) | 0 | 4
Ureteric stenosis (Renal and urinary disorders) | 1 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Urogenital fistula (Renal and urinary disorders) | 0 | 1
Vesicocutaneous fistula (Renal and urinary disorders) | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 2
Uterine fistula (Reproductive system and breast disorders) | 0 | 1
Vaginal fistula (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal ulceration (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Catheter placement (Surgical and medical procedures) | 1 | 0
Central venous catheter removal (Surgical and medical procedures) | 1 | 0
Chemotherapy (Surgical and medical procedures) | 1 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Cytoreductive surgery (Surgical and medical procedures) | 2 | 0
Ileostomy (Surgical and medical procedures) | 0 | 1
Intestinal resection (Surgical and medical procedures) | 0 | 1
Laparotomy (Surgical and medical procedures) | 0 | 2
Large intestine anastomosis (Surgical and medical procedures) | 0 | 1
Vaginal operation (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 4
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 5
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 4
Lymphocele (Vascular disorders) | 2 | 6
Lymphoedema (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 6
Varicose vein (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=450) | Nintedanib (N=902)
Anaemia (Blood and lymphatic system disorders) | 129 | 317
Leukopenia (Blood and lymphatic system disorders) | 78 | 165
Neutropenia (Blood and lymphatic system disorders) | 203 | 419
Thrombocytopenia (Blood and lymphatic system disorders) | 87 | 301
Abdominal distension (Gastrointestinal disorders) | 20 | 55
Abdominal pain (Gastrointestinal disorders) | 111 | 281
Abdominal pain upper (Gastrointestinal disorders) | 58 | 125
Constipation (Gastrointestinal disorders) | 151 | 254
Diarrhoea (Gastrointestinal disorders) | 114 | 692
Dyspepsia (Gastrointestinal disorders) | 24 | 77
Flatulence (Gastrointestinal disorders) | 9 | 53
Nausea (Gastrointestinal disorders) | 231 | 583
Stomatitis (Gastrointestinal disorders) | 24 | 51
Vomiting (Gastrointestinal disorders) | 119 | 391
Asthenia (General disorders) | 65 | 163
Fatigue (General disorders) | 201 | 388
Mucosal inflammation (General disorders) | 30 | 62
Oedema peripheral (General disorders) | 47 | 48
Pain (General disorders) | 27 | 35
Pyrexia (General disorders) | 46 | 64
Drug hypersensitivity (Immune system disorders) | 21 | 58
Hypersensitivity (Immune system disorders) | 32 | 53
Cystitis (Infections and infestations) | 17 | 66
Nasopharyngitis (Infections and infestations) | 36 | 73
Urinary tract infection (Infections and infestations) | 50 | 131
Alanine aminotransferase increased (Investigations) | 49 | 259
Aspartate aminotransferase increased (Investigations) | 41 | 219
Blood alkaline phosphatase increased (Investigations) | 16 | 74
Haemoglobin decreased (Investigations) | 24 | 56
Neutrophil count decreased (Investigations) | 23 | 74
Platelet count decreased (Investigations) | 17 | 63
Decreased appetite (Metabolism and nutrition disorders) | 63 | 168
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 85
Hypomagnesaemia (Metabolism and nutrition disorders) | 25 | 92
Arthralgia (Musculoskeletal and connective tissue disorders) | 137 | 242
Back pain (Musculoskeletal and connective tissue disorders) | 54 | 83
Bone pain (Musculoskeletal and connective tissue disorders) | 39 | 62
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 29 | 56
Myalgia (Musculoskeletal and connective tissue disorders) | 107 | 201
Pain in extremity (Musculoskeletal and connective tissue disorders) | 56 | 95
Dizziness (Nervous system disorders) | 36 | 77
Dysgeusia (Nervous system disorders) | 37 | 126
Headache (Nervous system disorders) | 53 | 140
Neuropathy peripheral (Nervous system disorders) | 85 | 172
Paraesthesia (Nervous system disorders) | 64 | 100
Peripheral sensory neuropathy (Nervous system disorders) | 114 | 214
Polyneuropathy (Nervous system disorders) | 25 | 50
Anxiety (Psychiatric disorders) | 27 | 36
Depression (Psychiatric disorders) | 32 | 51
Insomnia (Psychiatric disorders) | 57 | 105
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 57
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 | 109
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 72
Alopecia (Skin and subcutaneous tissue disorders) | 278 | 519
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 44
Rash (Skin and subcutaneous tissue disorders) | 50 | 95
Hot flush (Vascular disorders) | 45 | 73
Hypertension (Vascular disorders) | 23 | 119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights